CLINICAL TRIAL: NCT02502409
Title: Natural History Study of Factor IX Treatment and Complications
Acronym: B-Natural
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Skane University Hospital (Other)
Collaborators: Indiana Hemophilia &Thrombosis Center, Inc. (Other); Bioverativ Therapeutics Inc. (Industry); Swedish Orphan Biovitrum (Industry)
Responsible Party: Principal Investigator, Sharyne M. Donfield, Ph.D., Principal Investigator, Data Coordinating Center, Rho, Inc., Skane University Hospital
Other Study IDs: B-Natural
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Factor IX Deficiency
Keywords: Hemophilia B; Hemophilia B with Inhibitors
MeSH Terms: conditions — Hemophilia B | interventions — Standard of Care; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, cells
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Standard care with blood and urine sample collection

SUMMARY:
This study will examine two groups of subjects with factor IX (FIX) deficiency: 1) those with a current or history of inhibitors to FIX, and; 2) groups of two or more affected brothers, with or without inhibitors. The overall goal is to characterize the study groups in terms of their medical history, their patterns of bleeding, their care, quality of life, and complications including the development of joint disease, inhibitory antibodies to FIX, use of immune tolerance induction (ITI) and outcome.

DETAILED DESCRIPTION:
Hemophilia B, FIX deficiency, is the second most common type of hemophilia, occurring in about one in 25,000 male births. This disease is in some ways more complex than hemophilia A, and is less well understood. Differences include a lower incidence and a greater risk of side effects to treatment, for example, allergic reactions and kidney disease. This study will examine two groups of subjects with FIX deficiency - those with a current or history of inhibitors to FIX, and groups of two or more affected brothers, with or without inhibitors. The overall goal is to characterize the study group in terms of their medical history, their patterns of bleeding, their care, quality of life, and complications including the development of inhibitory antibodies to FIX, allergies, kidney, and joint disease.

ELIGIBILITY:
Inclusion Criteria:

1. A consent approved by the appropriate Institutional Review Board (IRB)/Independent Ethics Committee (IEC) has been obtained from the subject or his legally acceptable representative
2. Subject has FIX deficiency AND

   * Is part of an affected brother pair/group that will also enroll; AND/OR
   * Has a current or history of inhibitor, defined as >0.6 Bethesda units (BU)

Exclusion Criteria:

1. Subject has another congenital bleeding disorder
2. Subject is a carrier of hemophilia B with factor level >0.40 IU/mL

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population includes groups of two or more affected brothers, with or without a history of inhibitors, who share(d) one or both biological parents; and individuals with a history of an inhibitor. Most affected brother pairs will be concordant for no inhibitor and will serve as a control group for those with inhibitors. The study is open to subjects with mild (0.05-0.40 IU/mL), moderate (0.01-<0.05 IU/mL), or severe (<0.01 IU/mL) FIX deficiency. Females meeting the eligibility criteria may participate. There are no lower or upper age limits. Type of treatment, regimen, dosing and product(s) used are at the discretion of the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-06 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Inhibitory antibodies | Baseline
  Current or history of inhibitors
Annualized bleeding rate | 6 months
  Overall and by bleeding site
Joint assessment | Baseline
  Range of motion
Renal disorders | 6 months
  Reported subject and family history of renal disease
Hemophilia treatment adherence | Baseline
  Validated Hemophilia Regimen Treatment Adherence Scale--Prophylaxis (VERITAS-Pro), Validated Hemophilia Regimen Treatment Adherence Scale - PRN (VERITAS-PRN)
Health related quality of life | Baseline
  European Quality of Life - 5 Dimensions (EQ5D)
Non-inhibitory antibodies | Baseline
  Measured at central laboratory

SECONDARY OUTCOMES:
Factor IX usage | 6 months
  Treatment history with FIX replacement
Number of hospitalizations | 6 months
  Hospitalizations reported during 6 month follow up period
Number of surgical procedures | 6 months
  Surgical procedures reported during 6 month follow up period
number of days missed from school or work | 6 months
  Days missed from school or work during 6 month follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Erik Berntorp, MD, PhD, Study Director — Skåne University Hospital, Malmö; Amy D Shapiro, MD, Study Director — Indiana Hemophilia &Thrombosis Center, Inc.; Jan Astermark, MD, PhD, Study Director — Skåne University Hospital, Malmö; Christine Knoll, MD, Principal Investigator — Phoenix Children's Hospital, Phoenix, AZ; Yasmina Abajas, MD, Principal Investigator — University of North Carolina Hemophilia Treatment Center, Chapel Hill, NC; Catherine McGuinn, MD, Principal Investigator — Weill Cornell Medical College, New York, NY; Munira Borhany, MD, Principal Investigator — National Institute of Blood Disease and Bone Marrow Transplantation, Karachi, Pakistan; Philip Kuriakose, MD, Principal Investigator — Henry Ford Health System, Detroit, MI; Eva Funding, MD, Principal Investigator — National University Hospital Copenhagen, Copenhagen, Denmark; Stacy Croteau, MD, Principal Investigator — Boston Hemophilia Center, Boston, MA; Christine Kempton, MD, Principal Investigator — Emory University, Atlanta, Georgia; Susan Kearney, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota, Minneapolis, MN; Suchitra Acharya, MD, Principal Investigator — Cohen Children's Medical Center, New Hyde Park, NY; Roshni Kulkarni, MD, Principal Investigator — Michigan State University, East Lansing, MI; Raina Liesner, MD, Principal Investigator — Great Ormond Street Hospital for Children, London, UK; Christoph Bidlingmaier, MD, Principal Investigator — Dr. v Hauner Children's University Hospital, Munich, Germany; Alice J. Cohen, MD, Principal Investigator — Newark Beth Israel Medical Center, Newark, NJ; Manuela Carvalho, MD, Principal Investigator — Centro Hospitalar de São João, Porto, Portugal; Margaret Ragni, MD, Principal Investigator — University of Pittsburgh and Hemophilia Center of Western Pennsylvania, Pittburgh, PA US; Ulrike Reiss, MD, Principal Investigator — St. Jude Children's Research Hospital, Memphis, TN US; Michelle Witkop, DNP, FNP-BC, Principal Investigator — Munson Medical Center, Traverse City, MI, US; Katharina Holstein, MD, Principal Investigator — University Medical Centre Hamburg-Eppendorf, Hamburg, Germany; Cristina Tarango, MD, Principal Investigator — Cincinnati Children's Hospital Medical Center, Cincinnati, OH US; Michael D Tarantino, MD, Principal Investigator — Bleeding and Clotting Disorders Institute, Peoria, IL US; Johannes Oldenburg, MD, Ph.D, Principal Investigator — University Clinic, Bonn
Locations (1):
- Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Shapiro AD, Ragni MV, Borhany M, Abajas YL, Tarantino MD, Holstein K, Croteau SE, Liesner R, Tarango C, Carvalho M, McGuinn C, Funding E, Kempton CL, Bidlingmaier C, Cohen A, Oldenburg J, Kearney S, Knoll C, Kuriakose P, Acharya S, Reiss UM, Kulkarni R, Witkop M, Lethagen S, Donfield S, LeBeau P, Berntorp E, Astermark J. Natural history study of factor IX deficiency with focus on treatment and complications (B-Natural). Haemophilia. 2021 Jan;27(1):49-59. doi: 10.1111/hae.14139. Epub 2020 Dec 5. PMID 33278853